CLINICAL TRIAL: NCT01864213
Title: The Efficacy of Topical Amethocaine Gel in Reducing the Pain of Local Anesthetic Infiltration Prior to Neuraxial Anesthesia in Non-labouring Pregnant Women: A Randomized Controlled Trial
Brief Title: Efficacy of Ametop Cream in Reducing Pain of Local Anesthetic Infiltration
Acronym: Ametop
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: H13-00771
Record Dates: First submitted 2013-05-09; First posted 2013-05-29 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Tetracaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ametop cream (Experimental)
  Interventions: Drug: Ametop cream

INTERVENTIONS:
Drug: Ametop cream
  Other Names: amethocaine

SUMMARY:
Ametop is a numbing cream used to ease the pain of having blood drawn or an IV inserted. It is safe and virtually none enters the blood stream. It's effectiveness at reducing the pain of the freezing injection prior to epidural/ spinal anesthesia in pregnant women has not been studied.

DETAILED DESCRIPTION:
We propose to randomize 70 women to have either the numbing cream or a similar looking moisturizing cream placed on their lower back before their anesthetic. They will rate the discomfort of the freezing injection allowing us to compare the two groups and determine if the numbing cream is effective.

ELIGIBILITY:
Inclusion Criteria:

* Any pregnant subject undergoing an elective procedure under neuraxial anesthesia.

Exclusion Criteria:

* Any contraindication to neuraxial anesthesia
* Subjects in labour

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Pain score | Within 5 minutes of spinal
  Patient will be asked to give a pain score

CONTACTS AND LOCATIONS:
Overall Officials: Vit Gunka, MD FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada